CLINICAL TRIAL: NCT02708433
Title: Pilot Study: Comparison of Buffered 1% vs. Non-Buffered 2% Lidocaine Used in Dental and Oral Surgical Procedures: Clinical Outcomes
Brief Title: Clinical Outcomes of Buffered 1% Lidocaine vs. Non-buffered 2% Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-0068a
Record Dates: First submitted 2016-03-03; First posted 2016-03-15 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2017-10

CONDITIONS: Anesthesia
Keywords: lidocaine, jaw
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Buffered 1% lidocaine (Active Comparator): In week one each subject would receive either anesthetic (Buffered 1% lidocaine with 1/100,000 Epinephrine) or (Non-Buffered 2% lidocaine with 1/100,000 Epinephrine) to block the inferior alveolar, lingual, buccal nerves.
  In week two the alternate anesthetic would be administered.
  Mandibular molar and canine tested for pulpal anesthesia
  Interventions: Drug: Lidocaine
- Non-Buffered lidocaine (Active Comparator): In week two each subject would receive the alternate anesthetic (Buffered 1% lidocaine with 1/100,000 Epinephrine) or (Non-Buffered 2% lidocaine with 1/100,000 Epinephrine) to block the inferior alveolar, lingual, buccal nerves.
  Mandibular molar and canine tested for pulpal anesthesia
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine
  Other Names: xylocaine

SUMMARY:
Anecdotal data suggest that the buffered form of the local anesthetic is more potent at equal dosages, and a lower dosage of the drug might be used with an effect equal to higher dosage not buffered. Clinical data are needed to confirm these anecdotal data. No data exist comparing buffered local anesthetics at lower drug concentrations to current dosages commonly used in dental and oral surgical procedures

DETAILED DESCRIPTION:
Specific Aims:

Compare clinical depths of pulpal anesthesia (cold, Electronic Pulp Test) for mandibular molar, and canine teeth at 30 minute intervals post injection for mandibular block anesthesia with buffered 1% lidocaine with 1/100,000 epinephrine as compared to non-buffered 2% lidocaine with 1/100,000 epinephrine.

Hypotheses:

No differences exist in anesthetic depth for pulpal anesthesia after intraoral injection for mandibular block anesthesia between buffered 1% lidocaine with 1/100,000 epinephrine as compared to non-buffered 2% lidocaine with 1/100,000 epinephrine.

Study Time Frame: 6 months Month One: Recruit 24 volunteers as subjects. Prepare case-books. Months Two-Three: Clinical Study, Months Four-Five: Analyze data Month Six: Prepare Abstracts, Papers Methods: Blinded, Randomized Clinical Design Recruit subjects with Institutional Review Board approved consent at UNC Subjects will serve as their own controls in a cross-over AB/BA study design which is uniform within sequences, uniform within periods, and balanced Randomized subjects to be injected orally for mandibular block (inferior alveolar, lingual, buccal nerves) alternatively with 4cc of buffered 1% lidocaine with 1/100,000 epinephrine and 4cc non-buffered of 2% lidocaine with 1/100,000 epinephrine.

Assessment: pre, and post-anesthetic administration for pulpal anesthesia with cold, Electronic Pulp Test: Mandibular molar, canine at 30 minute intervals Inclusion Criteria: Age 18-30 years, American Society Anesthesiologists (ASA) I Exclusion Criteria Allergy to lidocaine class of anesthetic drugs, Local anesthetic drug past week Current symptoms teeth or oral mucosa. SAS will be used for database management and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years, ASA I

Exclusion Criteria:

* Allergy to lidocaine class of anesthetic drugs Local anesthetic drug use in past week Current symptoms teeth or oral mucosa

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P White, Jr., DDS, PhD, Principal Investigator — UNC Dept Oral and Maxillofacial Surgery
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine: At each treatment visit, participants were injected orally for mandibular block (inferior alveolar, lingual, buccal nerves).
  For this arm, participants first received Buffered 1% Lidocaine followed by a 1-week washout, then Non-buffered 2% Lidocaine.
- Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine: At each treatment visit, participants were injected orally for mandibular block (inferior alveolar, lingual, buccal nerves).
  For this arm, participants first received Non-Buffered 2% Lidocaine followed by a 1-week washout, then Buffered 1% Lidocaine.
Period: First Intervention (Visit 1)
Arm/Group | Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Washout (at Least 1 Week)
Arm/Group | Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Second Intervention (Visit 2)
Arm/Group | Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who were randomized to received either Buffered 1% Lidocaine or Non-buffered 2% Lidocaine
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Pulpal Response After Mandibular Molar Anesthesia
Description: Subject's Mandibular first molar teeth tested before anesthetic and every 30 minutes after for response to Cold and Electric Pulp Test as reported by subjects as a "yes" or "no."
Time Frame: Every 30 minutes up to 120 minutes total
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Number analyzed (Participants) | 23 | 23
Minutes | 99 (49) | 98 (45)
Statistical Analysis 1: Comparison: Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine vs Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine; Test type: Superiority; p = 0.74, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.49 to 0.57], Standard Deviation 49

2. Primary Outcome: Mean Time to Pulpal Response After Mandibular Canine Anesthesia
Description: Subject's Mandibular canine teeth will be tested before anesthetic and every 30 minutes after for response to Cold and Electronic Pulp Test for presence of anesthesia as reported by participants "yes" or "no."
Time Frame: Every 30 minutes up to 120 minutes total
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine | Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine
Number analyzed (Participants) | 23 | 23
Minutes | 82 (48) | 85 (48)
Statistical Analysis 1: Comparison: Buffered 1% Lidocaine, Then Non-buffered 2% Lidocaine vs Non-Buffered 2% Lidocaine, Then Buffered 1% Lidocaine; Test type: Superiority; p = 0.5, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.89 to 0.52], Standard Deviation 48

ADVERSE EVENTS:
Time Frame: Adverse events collected for 24 hours after active component of the trial
Groups:
- Buffered 1% Lidocaine: At each treatment visit, participants were injected orally for mandibular block (inferior alveolar, lingual, buccal nerves).
  For this arm, participants first received Buffered 1% Lidocaine followed by a 1-week washout, then Non-buffered 2% Lidocaine.
- Non-Buffered 2% Lidocaine: At each treatment visit, participants were injected orally for mandibular block (inferior alveolar, lingual, buccal nerves).
  For this arm, participants first received Non-Buffered 2% Lidocaine followed by a 1-week washout, then Buffered 1% Lidocaine.
Arm/Group | Buffered 1% Lidocaine | Non-Buffered 2% Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02708433/Prot_SAP_000.pdf